CLINICAL TRIAL: NCT00809315
Title: Intervention Development and Pilot for Foster Care Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Kempe Foundation for the Prevention and Treatment of Child Abuse and Neglect (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 02-0516a; R21MH067618 (NIH)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Child Abuse
Keywords: Child abuse and neglect; Out-of-home care; Mentoring; Skills groups; Assessment; Functioning as a result of maltreatment and placement in out-of-home care
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assessment only (Active Comparator): Cognitive, academic achievement and mental health screening assessment and report.
  Interventions: Other: Assessment
- Fostering Healthy Futures (FHF) Assessment + FHF (Experimental): Cognitive, academic achievement and mental health screening assessment and report. Weekly therapeutic skill groups and mentoring over a 9-month period.
  Interventions: Other: Assessment; Behavioral: Fostering Healthy Futures (FHF)

INTERVENTIONS:
Other: Assessment — Cognitive, academic achievement, and mental health screening assessment and report.
Behavioral: Fostering Healthy Futures (FHF) — Weekly therapeutic skill groups and mentoring over a 9-month period.
  Arms: Fostering Healthy Futures (FHF) Assessment + FHF

SUMMARY:
The purpose of this study is to develop, standardize and provide a preliminary test of a novel intervention for preadolescent maltreated youth in out-of-home care. It is hypothesized that the preventive intervention, which is known as Fostering Healthy Futures (FHF) and which consists of therapeutic skills groups and mentoring, will improve mental health, social, academic and behavioral functioning and reduce youths' initiation of, and participation in, problem behaviors.

DETAILED DESCRIPTION:
This R21 application for a 3-year exploratory/development grant for intervention research is designed to develop, standardize and provide a preliminary test of a novel intervention for children, ages 9-11, placed in out-of-home care. Children and adolescents with a history of maltreatment and subsequent placement in foster care are at risk for substantial mental health and behavioral problems of great public health significance. In the prior longitudinal work with children in foster care, the investigators have described the population, examined child welfare system impact, and identified modifiable psychosocial risk and protective factors. These pre-intervention activities, supported by the principal investigator's K01 award, have enabled the investigator to address important methodological issues that have hampered the development of intervention efforts targeting this high-risk population.

Based on this pre-intervention research, feedback from focus group participants, and a review of other efficacious programs for high-risk youth, the investigators propose to design an intervention for preadolescent youth in foster care consisting of three primary components: assessment and advocacy, mentoring, and therapeutic skills groups. The proposed R21 activities include developing the assessment battery and intervention protocol, manualizing the treatment, estimating recruitment and attrition rates, and conducting a small-scale randomized-controlled pilot study of the intervention. The goals of the intervention will be to improve mental health, social, academic and behavioral functioning and to reduce youths' initiation of, and participation in, problem behaviors. The investigators will conduct a preliminary examination of whether these proximal outcomes are moderated by baseline characteristics and/or mediated by the process variables targeted by the intervention. Estimates of effect size will be used to determine the sample size needed for adequate power to conduct a full-scale randomized controlled trial. The pilot study will also focus on issues of feasibility, program uptake, and replicability, and the investigators will modify the assessment battery, protocol, and manuals following the pilot phase and prior to the application for an R01 to conduct a large-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

All of the 9-11-year-old children court-ordered into out-of-home care (as a result of maltreatment) over the prior year in participating counties, including:

1. Youth placed in group homes, foster homes, and with kin
2. Youth with significant behavior problems
3. Youth who meet criteria for mental health diagnoses or dual diagnosis
4. Youth with mild cognitive impairment

Exclusion Criteria:

1. Youth who reunify before the beginning of the intervention
2. Youth with significant cognitive, behavioral, and/or mental health impairment that interfered with either with their ability to benefit from the prevention program or to participate safely
3. Youth who were not proficient enough in English to participate
4. Youth who lived too far from sites where groups were hel

When siblings were both eligible, only one sibling was randomly selected to participate in the study, and the other(s) was excluded

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2002-08; Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of Child mental health, social & behavioral functioning and quality of life as measured from multiple informants and sources. | Immediately post-intervention and 6-months post intervention

SECONDARY OUTCOMES:
Evaluation of Problem behaviors, life-course outcomes, placement history, and service system involvement as measured from multiple informants and sources. | Immediately post-intervention, 6-months post-intervention, 2.5 years post-intervention and possible future timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Heather N Taussig, PhD, Principal Investigator — University of Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Taussig HN, Culhane SE, Hettleman D. Fostering healthy futures: an innovative preventive intervention for preadolescent youth in out-of-home care. Child Welfare. 2007 Sep-Oct;86(5):113-31. PMID 18422051
- [Result] Taussig HN, Culhane SE. Impact of a mentoring and skills group program on mental health outcomes for maltreated children in foster care. Arch Pediatr Adolesc Med. 2010 Aug;164(8):739-46. doi: 10.1001/archpediatrics.2010.124. PMID 20679165
- [Result] Taussig HN, Culhane SE, Garrido E, Knudtson MD. RCT of a mentoring and skills group program: placement and permanency outcomes for foster youth. Pediatrics. 2012 Jul;130(1):e33-9. doi: 10.1542/peds.2011-3447. Epub 2012 Jun 11. PMID 22689870
- [Derived] Hambrick E, Lee SK, Weiler L, Collins JO, Rhodes T, Taussig H. Engagement in a Preventive Intervention for Preadolescent Children in Foster Care: Considerations for Intervention Design. Child Psychiatry Hum Dev. 2023 Oct;54(5):1373-1385. doi: 10.1007/s10578-022-01341-8. Epub 2022 Mar 18. PMID 35303199
- [Derived] Taussig HN, Dmitrieva J, Garrido EF, Cooley JL, Crites E. Fostering Healthy Futures Preventive Intervention for Children in Foster Care: Long-term Delinquency Outcomes from a Randomized Controlled Trial. Prev Sci. 2021 Nov;22(8):1120-1133. doi: 10.1007/s11121-021-01235-6. Epub 2021 Apr 27. PMID 33905053